CLINICAL TRIAL: NCT06139757
Title: Sleep Length and Euploid Embryo Transfer Prospective Study
Acronym: SLEEP
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Friends of Prentice (Other)
Responsible Party: Principal Investigator, Jessica Walter, Professor, Northwestern University
Other Study IDs: STU00219133
Record Dates: First submitted 2023-10-28; First posted 2023-11-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female
Keywords: wearable; sleep
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Euploid embryo transfer group: Participants will wear the Oura Ring continuously for data collection starting in the month prior to their embryo transfer date. They will wear the Oura Ring throughout the preparation, embryo transfer, and post-transfer until either a negative pregnancy test or, if positive, until 8 weeks gestation. The study time for each participant will thus extend from either 5 weeks for negative pregnancy tests, to 10 weeks for normally continuing pregnancies.
  Interventions: Device: Oura ring

INTERVENTIONS:
Device: Oura ring — Patient will wear Oura ring before and after embryo transfer. They will be blinded to sleep data during this period. Thus the intervention of wearing the ring to track sleep will not affect outcomes, but rather track the outcome of sleep.

SUMMARY:
Sleep is a critical component of daily life that significantly influences health and well-being. Despite the integral role sleep plays in life, its effect on women's reproductive health, and its subsequent impact on fertility, is largely understudied. The purpose of the SLEEP Study is to investigate the link between sleep and fertility. Participants will use a wireless wearable device mounted on the finger to measure sleep in the weeks preceding and following an embryo transfer during treatment with in vitro fertilization. The investigators hope that these findings will inform future therapies that improve sleep and fertility outcomes.

DETAILED DESCRIPTION:
Infertility is a devastating disease affecting 1 in 8 couples in the United States and over 80 million people worldwide. Despite significant improvements in the treatments available to infertile individuals in recent decades, there is a high dropout rate due to treatment cost, and treatment success is variable. Even in the setting of a genetically normal embryo, live birth rates after chromosomally normal (i.e. euploid) embryo transfers hover around 60%. Infertility is also associated with significant morbidities among those affected, ranging from emotional suffering, anxiety and depression, to overwhelming financial burden and isolating social stigma.

Although the underlying etiologies of infertility vary greatly, a common denominator shared by a disproportionate number of infertile women is poor sleep. Physicians routinely screen for diabetes and thyroid disease, yet rarely consider the contribution of sleep to healthy reproductive outcomes. This is partially due to the challenges with studying, measuring and quantifying sleep. However, with the advent of commercially available wearable devices, the scientific community has a new and exciting opportunity to quantify the potential harm of poor sleep and identify a new treatment avenue for infertile couples.

Sleep is a critical component of daily life that significantly influences health and well-being. On average, humans spend one third of life asleep. Yet, with the increasing pressures toward high-productivity, and that demand slowly turning us into a '24-hour society,' many Americans are becoming chronically under slept in the last several decades. Recent estimates purport that over 1 in 3 people in the U.S. sleep less than the recommended minimum of 7 hours a night. Among women of reproductive age, a similarly large group has chronic sleep deficits, with approximately 30% of women self-reporting no more than 6 hours of nightly sleep. Poor sleep quality has been linked to multiple co-morbidities, including anxiety, depression, obesity, diabetes, hypertension, myocardial infarct, and stroke. Moreover, deficits in the most important stage of sleep known as rapid-eye-movement (REM) sleep, have been linked to increased mortality and cognitive decline. Thus, sleep represents an important modifiable risk factor in human well and disease states across the lifespan.

Despite the integral role sleep plays in life, its effect on women's reproductive health, and its subsequent impact on fertility, is largely understudied. Animal models of disrupted sleep have shown significant effects of circadian rhythm alterations on reproductive hormone function, leading to both ovulatory dysfunction and sub-fertility. A murine knock-out model of certain circadian rhythm genes (known as 'Clock' genes) found lower rates of embryo implantation due to decreased steroid hormone production. Human subjects research has largely focused on night-shift workers as a model for abnormal sleep. Women in this group have demonstrated higher rates of irregular menstrual cycles and infertility. Moreover, women with circadian disruption due to working at night had increased rates of pregnancy loss compared to women working during the day. Even among women with night-time sleeping schedules, less sleep has been noted as a risk factor for first and second trimester miscarriages. Based on these studies, sleep and circadian rhythms may play a role in both achieving and sustaining pregnancy.

While studies have shown high rates of both psychological distress and poor sleep among women presenting to fertility clinics, a direct link between sleep and fertility has yet to be demonstrated. This proposed study aims to investigate if this link exists, as understanding the relationship between a 'good night's sleep' and one's reproductive potential could inform future therapies to modify sleep as a risk factor and decrease rates of infertility in women across the lifespan.

There are few studies exploring the complex relationship between infertility, sleep, and reproductive outcomes. Prior studies relied on subjective measures of sleep (e.g. sleep diaries and questionnaires) to measure total sleep time prior to and after in vitro fertilization and embryo transfer. Self-reported sleep estimates are notoriously inaccurate and over-report total sleep time compared to polysomnography and actigraphy measures. Furthermore, only one study used actigraphy, a non-invasive, wrist-mounted device, to objectively measure sleep, but was limited by a small sample size and use of surrogate measures of success (e.g. number of oocytes retrieved and embryos made during IVF), rather than pregnancy or live birth rates, compromising an ability to draw meaningful conclusions and implications for pregnancy rates.

This proposal will be the first adequately powered prospective study to comprehensively measure sleep quality and quantity prior to embryo transfer. Validated sleep questionnaires in combination with continuous actigraphy data collected by the Oura ring will be used, a finger-mounted multi-sensor sleep tracker that performs well compared to the gold-standard in sleep tracking of laboratory polysomnography. This study will prospectively follow participants from the 3-4 weeks preceding an embryo transfer, into the weeks following an embryo transfer and early pregnancy. Comprehensive and objective data generated by the Oura ring will be leveraged to characterize the effects of sleep on pregnancy outcomes.

The investigators hypothesize that lower average total sleep time in the month preceding a frozen embryo transfer will be associated with lower implantation, clinical pregnancy, and ongoing pregnancy rates after single euploid embryo transfers. The investigators further hypothesize that lower average total sleep time in the month after frozen euploid embryo transfer will be associated with higher rates of miscarriage. Secondary hypotheses will assess whether or not additional sleep parameters (sleep onset, wake time, sleep midpoint, amount of night time awakenings, and nighttime heart rate variability) are associated with the same positive or negative pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a single euploid frozen embryo transfer
* Patient's 1st, 2nd, or 3rd embryo transfer (prior fresh or frozen transfers included)

Exclusion Criteria:

* Primary infertility diagnosis of polycystic ovary syndrome
* BMI > 40
* Diagnosis of primary ovarian insufficiency (FSH > 40)
* Night work
* High risk of poor outcomes of fertility treatment [> 2 prior miscarriages (women with recurrent pregnancy loss), significant uterine factor infertility [>/= 2 myomectomies (open abdominal or laparoscopic) or any non-hystoeroscopic myomectomy entering the endometrial cavity]
* Undergoing medical fertility preservation for a significant medical co-morbidity
* Current cancer diagnosis
* > 3 prior failed embryo transfers in attempt for current live birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients anticipating frozen embryo transfer of a genetically tested, euploid embryo at Northwestern's Center for Fertility and Reproductive Medicine.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Effect of sleep on IVF outcomes | Sleep parameters will be measured on a daily basis
  To elucidate a potential correlation between average total sleep time and other sleep parameters (sleep efficiency, wake after sleep onset, and sleep stages) during the pre- and post-embryo transfer windows on rates of implantation, clinical pregnancy, ongoing pregnancy, and miscarriage.

SECONDARY OUTCOMES:
Effect of anxiety on sleep parameters | Anxiety will be assessed at baseline with GAD-7
  To analyze if there are any differences between sleep parameters in women with different fertility diagnoses, and varying levels of anxiety on a validated questionnaire.
Effect of depression on sleep parameters | Depressive symptoms will be assessed at baseline with PHQ-9
  To analyze if there are any differences between sleep parameters in women with different fertility diagnoses, and varying levels of depressed mood on a validated questionnaire
Effect of frozen embryo transfer protocol type on sleep parameters and pregnancy outcomes | Sleep parameters will be measured on a daily basis. Pregnancy outcomes will be measured at time of pregnancy testing, and if positive up to 8-10 weeks of gestation
  To compare if there are sleep differences (total sleep time) and pregnancy outcome differences (implantation rate, live birth rate, miscarriage rate) in women undergoing a natural cycle frozen embryo transfer, which utilizes natural ovulation to time embryo transfer, compared to an artificial or medicated cycle frozen embryo transfer, wherein the natural menstrual cycle is suppressed and the uterine lining prepared for transfer using pharmacologic preparations of estrogen and progesterone.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Walter, MD, MSCE, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoma ME, McLain AC, Louis JF, King RB, Trumble AC, Sundaram R, Buck Louis GM. Prevalence of infertility in the United States as estimated by the current duration approach and a traditional constructed approach. Fertil Steril. 2013 Apr;99(5):1324-1331.e1. doi: 10.1016/j.fertnstert.2012.11.037. Epub 2013 Jan 3. PMID 23290741
- [Background] Cousineau TM, Domar AD. Psychological impact of infertility. Best Pract Res Clin Obstet Gynaecol. 2007 Apr;21(2):293-308. doi: 10.1016/j.bpobgyn.2006.12.003. Epub 2007 Jan 22. PMID 17241818
- [Background] Eryilmaz OG, Devran A, Sarikaya E, Aksakal FN, Mollamahmutoglu L, Cicek N. Melatonin improves the oocyte and the embryo in IVF patients with sleep disturbances, but does not improve the sleeping problems. J Assist Reprod Genet. 2011 Sep;28(9):815-20. doi: 10.1007/s10815-011-9604-y. Epub 2011 Jul 12. PMID 21748445
- [Background] Ford ES, Cunningham TJ, Croft JB. Trends in Self-Reported Sleep Duration among US Adults from 1985 to 2012. Sleep. 2015 May 1;38(5):829-32. doi: 10.5665/sleep.4684. PMID 25669182
- [Background] Beroukhim G, Esencan E, Seifer DB. Impact of sleep patterns upon female neuroendocrinology and reproductive outcomes: a comprehensive review. Reprod Biol Endocrinol. 2022 Jan 18;20(1):16. doi: 10.1186/s12958-022-00889-3. PMID 35042515
- [Background] Consensus Conference Panel; Watson NF, Badr MS, Belenky G, Bliwise DL, Buxton OM, Buysse D, Dinges DF, Gangwisch J, Grandner MA, Kushida C, Malhotra RK, Martin JL, Patel SR, Quan SF, Tasali E. Joint Consensus Statement of the American Academy of Sleep Medicine and Sleep Research Society on the Recommended Amount of Sleep for a Healthy Adult: Methodology and Discussion. Sleep. 2015 Aug 1;38(8):1161-83. doi: 10.5665/sleep.4886. PMID 26194576
- [Background] White ND. Influence of Sleep on Fertility in Women. Am J Lifestyle Med. 2016 Apr 3;10(4):239-241. doi: 10.1177/1559827616641386. eCollection 2016 Jul-Aug. PMID 30202278
- [Background] Worley SL. The Extraordinary Importance of Sleep: The Detrimental Effects of Inadequate Sleep on Health and Public Safety Drive an Explosion of Sleep Research. P T. 2018 Dec;43(12):758-763. PMID 30559589
- [Background] Leary EB, Watson KT, Ancoli-Israel S, Redline S, Yaffe K, Ravelo LA, Peppard PE, Zou J, Goodman SN, Mignot E, Stone KL. Association of Rapid Eye Movement Sleep With Mortality in Middle-aged and Older Adults. JAMA Neurol. 2020 Oct 1;77(10):1241-1251. doi: 10.1001/jamaneurol.2020.2108. PMID 32628261
- [Background] Suh SW, Han JW, Lee JR, Byun S, Kwak KP, Kim BJ, Kim SG, Kim JL, Kim TH, Ryu SH, Moon SW, Park JH, Seo J, Youn JC, Lee DY, Lee DW, Lee SB, Lee JJ, Jhoo JH, Yoon IY, Kim KW. Short Average Duration of NREM/REM Cycle Is Related to Cognitive Decline in an Elderly Cohort: An Exploratory Investigation. J Alzheimers Dis. 2019;70(4):1123-1132. doi: 10.3233/JAD-190399. PMID 31322573
- [Background] Sciarra F, Franceschini E, Campolo F, Gianfrilli D, Pallotti F, Paoli D, Isidori AM, Venneri MA. Disruption of Circadian Rhythms: A Crucial Factor in the Etiology of Infertility. Int J Mol Sci. 2020 May 30;21(11):3943. doi: 10.3390/ijms21113943. PMID 32486326
- [Background] Sen A, Hoffmann HM. Role of core circadian clock genes in hormone release and target tissue sensitivity in the reproductive axis. Mol Cell Endocrinol. 2020 Feb 5;501:110655. doi: 10.1016/j.mce.2019.110655. Epub 2019 Nov 19. PMID 31756424
- [Background] Ratajczak CK, Boehle KL, Muglia LJ. Impaired steroidogenesis and implantation failure in Bmal1-/- mice. Endocrinology. 2009 Apr;150(4):1879-85. doi: 10.1210/en.2008-1021. Epub 2008 Dec 4. PMID 19056819
- [Background] Ahlborg G Jr, Axelsson G, Bodin L. Shift work, nitrous oxide exposure and subfertility among Swedish midwives. Int J Epidemiol. 1996 Aug;25(4):783-90. doi: 10.1093/ije/25.4.783. PMID 8921457
- [Background] Stocker LJ, Macklon NS, Cheong YC, Bewley SJ. Influence of shift work on early reproductive outcomes: a systematic review and meta-analysis. Obstet Gynecol. 2014 Jul;124(1):99-110. doi: 10.1097/AOG.0000000000000321. PMID 24901274
- [Background] Infante-Rivard C, David M, Gauthier R, Rivard GE. Pregnancy loss and work schedule during pregnancy. Epidemiology. 1993 Jan;4(1):73-5. doi: 10.1097/00001648-199301000-00013. PMID 8420585
- [Background] Grajewski B, Whelan EA, Lawson CC, Hein MJ, Waters MA, Anderson JL, MacDonald LA, Mertens CJ, Tseng CY, Cassinelli RT 2nd, Luo L. Miscarriage among flight attendants. Epidemiology. 2015 Mar;26(2):192-203. doi: 10.1097/EDE.0000000000000225. PMID 25563432
- [Background] Samaraweera Y, Abeysena C. Maternal sleep deprivation, sedentary lifestyle and cooking smoke: Risk factors for miscarriage: A case control study. Aust N Z J Obstet Gynaecol. 2010 Aug;50(4):352-7. doi: 10.1111/j.1479-828X.2010.01190.x. PMID 20716263
- [Background] Philipsen MT, Knudsen UB, Zachariae R, Ingerslev HJ, Hvidt JEM, Frederiksen Y. Sleep, psychological distress, and clinical pregnancy outcome in women and their partners undergoing in vitro or intracytoplasmic sperm injection fertility treatment. Sleep Health. 2022 Apr;8(2):242-248. doi: 10.1016/j.sleh.2021.10.011. Epub 2021 Dec 20. PMID 34949542
- [Background] Yao QY, Yuan XQ, Liu C, Du YY, Yao YC, Wu LJ, Jiang HH, Deng TR, Guo N, Deng YL, Zeng Q, Li YF. Associations of sleep characteristics with outcomes of IVF/ICSI treatment: a prospective cohort study. Hum Reprod. 2022 May 30;37(6):1297-1310. doi: 10.1093/humrep/deac040. PMID 35259255
- [Background] Reschini M, Buoli M, Facchin F, Limena A, Dallagiovanna C, Bollati V, Somigliana E. Women's quality of sleep and in vitro fertilization success. Sci Rep. 2022 Oct 19;12(1):17477. doi: 10.1038/s41598-022-22534-0. PMID 36261696
- [Background] Lauderdale DS, Knutson KL, Yan LL, Liu K, Rathouz PJ. Self-reported and measured sleep duration: how similar are they? Epidemiology. 2008 Nov;19(6):838-45. doi: 10.1097/EDE.0b013e318187a7b0. PMID 18854708
- [Background] Matthews KA, Patel SR, Pantesco EJ, Buysse DJ, Kamarck TW, Lee L, Hall MH. Similarities and differences in estimates of sleep duration by polysomnography, actigraphy, diary, and self-reported habitual sleep in a community sample. Sleep Health. 2018 Feb;4(1):96-103. doi: 10.1016/j.sleh.2017.10.011. Epub 2017 Dec 13. PMID 29332687
- [Background] de Zambotti M, Cellini N, Menghini L, Sarlo M, Baker FC. Sensors Capabilities, Performance, and Use of Consumer Sleep Technology. Sleep Med Clin. 2020 Mar;15(1):1-30. doi: 10.1016/j.jsmc.2019.11.003. Epub 2020 Jan 3. PMID 32005346
- [Background] Goldstein CA, Lanham MS, Smith YR, O'Brien LM. Sleep in women undergoing in vitro fertilization: a pilot study. Sleep Med. 2017 Apr;32:105-113. doi: 10.1016/j.sleep.2016.12.007. Epub 2016 Dec 21. PMID 28366321
- [Background] Altini M, Kinnunen H. The Promise of Sleep: A Multi-Sensor Approach for Accurate Sleep Stage Detection Using the Oura Ring. Sensors (Basel). 2021 Jun 23;21(13):4302. doi: 10.3390/s21134302. PMID 34201861
- [Background] Miller DJ, Sargent C, Roach GD. A Validation of Six Wearable Devices for Estimating Sleep, Heart Rate and Heart Rate Variability in Healthy Adults. Sensors (Basel). 2022 Aug 22;22(16):6317. doi: 10.3390/s22166317. PMID 36016077
- [Background] Kocevska D, Lysen TS, Dotinga A, Koopman-Verhoeff ME, Luijk MPCM, Antypa N, Biermasz NR, Blokstra A, Brug J, Burk WJ, Comijs HC, Corpeleijn E, Dashti HS, de Bruin EJ, de Graaf R, Derks IPM, Dewald-Kaufmann JF, Elders PJM, Gemke RJBJ, Grievink L, Hale L, Hartman CA, Heijnen CJ, Huisman M, Huss A, Ikram MA, Jones SE, Velderman MK, Koning M, Meijer AM, Meijer K, Noordam R, Oldehinkel AJ, Groeniger JO, Penninx BWJH, Picavet HSJ, Pieters S, Reijneveld SA, Reitz E, Renders CM, Rodenburg G, Rutters F, Smith MC, Singh AS, Snijder MB, Stronks K, Ten Have M, Twisk JWR, Van de Mheen D, van der Ende J, van der Heijden KB, van der Velden PG, van Lenthe FJ, van Litsenburg RRL, van Oostrom SH, van Schalkwijk FJ, Sheehan CM, Verheij RA, Verhulst FC, Vermeulen MCM, Vermeulen RCH, Verschuren WMM, Vrijkotte TGM, Wijga AH, Willemen AM, Ter Wolbeek M, Wood AR, Xerxa Y, Bramer WM, Franco OH, Luik AI, Van Someren EJW, Tiemeier H. Sleep characteristics across the lifespan in 1.1 million people from the Netherlands, United Kingdom and United States: a systematic review and meta-analysis. Nat Hum Behav. 2021 Jan;5(1):113-122. doi: 10.1038/s41562-020-00965-x. Epub 2020 Nov 16. PMID 33199855
- [Background] Roehrs T, Kapke A, Roth T, Breslau N. Sex differences in the polysomnographic sleep of young adults: a community-based study. Sleep Med. 2006 Jan;7(1):49-53. doi: 10.1016/j.sleep.2005.05.008. Epub 2005 Sep 27. PMID 16194623
- [Background] Moraes W, Piovezan R, Poyares D, Bittencourt LR, Santos-Silva R, Tufik S. Effects of aging on sleep structure throughout adulthood: a population-based study. Sleep Med. 2014 Apr;15(4):401-9. doi: 10.1016/j.sleep.2013.11.791. Epub 2014 Feb 26. PMID 24657204
- [Background] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942
- [Background] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996
- [Background] Liu Z, Zheng Y, Wang B, Li J, Qin L, Li X, Liu X, Bian Y, Chen Z, Zhao H, Zhao S. The impact of sleep on in vitro fertilization embryo transfer outcomes: a prospective study. Fertil Steril. 2023 Jan;119(1):47-55. doi: 10.1016/j.fertnstert.2022.10.015. Epub 2022 Nov 23. PMID 36435629
- [Background] Roberts DM, Schade MM, Mathew GM, Gartenberg D, Buxton OM. Detecting sleep using heart rate and motion data from multisensor consumer-grade wearables, relative to wrist actigraphy and polysomnography. Sleep. 2020 Jul 13;43(7):zsaa045. doi: 10.1093/sleep/zsaa045. PMID 32215550
- [Background] Stone JD, Rentz LE, Forsey J, Ramadan J, Markwald RR, Finomore VS, Galster SM, Rezai A, Hagen JA. Evaluations of Commercial Sleep Technologies for Objective Monitoring During Routine Sleeping Conditions. Nat Sci Sleep. 2020 Oct 27;12:821-842. doi: 10.2147/NSS.S270705. eCollection 2020. PMID 33149712
- See also: World Health Organization. Current Practices and Controversies in Assisted Production. Geneva, Switzerland, 2002. — https://iris.who.int/bitstream/handle/10665/42576/9241590300.pdf?sequence=1
- See also: Sleep disturbances high in patients seeking fertility preservation — https://doi.org/10.1016/j.fertnstert.2013.07.1463